# School-based eHealth NCD Prevention Program to Improve Awareness in Adolescents from Urban Pakistan

**Document Date: 14- December- 2023** 

### **INFORMED CONSENT FORM**

### **INDEX**

| Pre Intervention | 3 |
|---|---|
| Focus Group Discussion | 3 |
| Assent Form for Pre-Intervention Focus Group Discussion of Students | 4 |
| Consent Form for Pre-Intervention Focus Group Discussion of Students from | Parents . 7 |
| Informed Consent for Pre-Intervention Focus Group Discussion of Teachers | 10 |
| Key Informant Interview | 13 |
| Informed Consent for Pre-Intervention Key Informant Interview - Administrat | ors 14 |
| Informed Consent for Pre-Intervention Key Informant Interview – Parent or G | uardian 17 |
| Intervention | 20 |
| Assent Form for Students for interventional study (School based eHealth NCD P | revention |
| Program) | 21 |
| Consent Form from Parents for their child participation in interventional study ( | School |
| based eHealth NCD Prevention Program) | 23 |
| Post Intervention | 26 |
| Assent Form for Post-Intervention Focus Group Discussion of Students | 27 |
| Consent Form for Post-Intervention Focus Group Discussion of Students | 30 |

## **Pre Intervention**

**Focus Group Discussion** 

# **Assent Form for Pre-Intervention Focus Group Discussion of Students**



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of<br>Health's Fogarty International Center<br>(FIC) in collaboration with Dept of<br>Medicine, Aga Khan University,<br>Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan<br>University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 1. Dr. Aysha Almas 2. Dr. Zainab Samad 3. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. PURPOSE OF THIS PROJECT

You have been invited to participate in a focus group discussion as part of the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors.

The purpose of the FGD is to explore participants' views regarding the barriers and facilitators associated with implementing the school-based eHealth NCD prevention program in schools. Furthermore, the participants' viewpoints on the content and design of the program will also be explored.

#### 2. PROCEDURES

The group discussion will be conducted at a secure and comfortable space within the school premises, such as a school library or study room with 6 to 8 other students. This discussion will be guided by your experiences, perceptions, and suggestions. A team of two members will conduct this discussion, one will moderate the session, and

the other will record the responses, both in writing and by audio recorder. The group discussion will take about 45 minutes

#### 3. POSSIBLE RISKS OR DISCOMFORT

We do not anticipate any risk or discomfort to you. However, you may decide not to respond to any probes if you feel they are too personal or if talking about them makes you uncomfortable.

#### 4. POSSIBLE BENEFITS

Your active participation in the group discussions will enable us to gain insights into your perspectives on the challenges and facilitators involved in implementing the School-based eHealth NCD prevention program in Pakistani schools. Additionally, these discussions will help us design and develop culturally tailored content for the video sessions and features of the eHealth application.

#### 5. FINANCIAL CONSIDERATIONS

You will be provided meal and travel allowance (if applicable) to participate in the FGD.

#### 6. CONFIDENTIALITY

All information that you provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your personal details. However, any information obtained as a result of your participation in the project may be inspected by the sponsor or by AKU ERC members.

#### 7. TERMINATION OF PROJECT

You are free to choose whether or not to participate in this project. There will be no penalty or loss of benefits to which you are otherwise entitled, if you choose not to participate.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### 9. AUTHORIZATION

I have read and understood this form, and I volunteer to participate in group-discussion as part of School-based eHealth NCD Prevention Program. I understand that I will receive a copy of this form. I voluntarily choose to participate, but I understand that my consent does not take away any legal rights in the case of negligence or other legal faults of anyone who is involved in this project.

| Name of participant (Printed or Typed): Date: |
|---------------------------------------------------|
| Signature/Thumb Impression of participant : Date: |
| Name of witness (Printed or Typed):<br>Date: |
| Signature/Thumb Impression of the witness: Date: |
| Signature of Principal/Co- Investigator:<br>Date: |
| Signature of the person obtaining consent: Date: |

### Consent Form for Pre-Intervention Focus Group Discussion of Students from Parents



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of<br>Health's Fogarty International Center<br>(FIC) in collaboration with Dept of<br>Medicine, Aga Khan University,<br>Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: Aga Khan University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 4. Dr. Aysha Almas 5. Dr. Zainab Samad 6. Muhammad Shahid Khan | Organization:<br>Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. Introduction

The purpose of this form is to provide you (as the parent of a prospective research study participant) information that may affect your decision as to whether or not to let your child participate in this research study. The person performing the research will describe the study to you and answer all your questions. Read the information below and ask any questions you might have before deciding whether or not to give your permission for your child to take part. If you decide to let your child participate in this study, this form will be used to record your permission.

#### 2. PURPOSE OF THIS PROJECT

If you agree, your child will be asked to participate in a focus group discussion as part of the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors. The purpose of the FGD is to explore participants' views regarding the barriers and facilitators associated with implementing the school-based eHealth NCD prevention program in schools. Furthermore, the participants' viewpoints on the content and design of the program will also be explored.

#### 3. PROCEDURES

The group discussion will be conducted at a secure and comfortable space within the school premises, such as a school library or study room with 6 to 8 other students. This discussion will be guided by your child's experiences, perceptions, and suggestions. A team of two members will conduct this discussion, one will moderate the session, and the other will record the responses, both in writing and by audio recorder. The group discussion will take about 45 minutes.

#### 4. POSSIBLE RISKS OR DISCOMFORT

We do not anticipate any risk or discomfort to the participant. However, your child may decide not to respond to any probes if s/he feel they are too personal or if talking about them makes him/her uncomfortable.

#### 5. POSSIBLE BENEFITS

Your child's active participation in the group discussions will enable us to gain insights on the challenges and facilitators involved in implementing the School-based eHealth NCD prevention program in Pakistani schools. Additionally, the discussion will help us design and develop culturally tailored content for the video sessions and features of the eHealth application.

#### 6. FINANCIAL CONSIDERATIONS

Your child will be provided meal and travel allowance (if applicable) to participate in the FGD.

#### 7. CONFIDENTIALITY

your child's privacy and the confidentiality of his/her data will be protected by keeping all information that your child provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your child's personal details. Your child's research records will not be released without your consent unless required by law or a court order. If it becomes necessary for the Ethics Review Committee to review the study records, information that can be linked to your child will be protected to the extent permitted by law. The data resulting from your child's participation may be made available to other researchers in the future for research purposes without identification. In these cases, the data will contain no identifying information that could associate it with your child, or with your child's participation in any study.

#### 8. TERMINATION OF PROJECT

You and your child's participation in this study is voluntary. Your child may decline to participate or to withdraw from participation at any time. Withdrawal or refusing to participate will not affect their treatment/procedure or relationship with Aga Khan University in anyway. You can agree to allow your child to be in the study now and change your mind later without any penalty.

In addition to your permission, your child must agree to participate in the study. If your child does not want to participate they will not be included in the study and there will be no penalty. If your child initially agrees to be in the study s/he can change their mind later without any penalty.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### **AUTHORIZATION**

You are making a decision about allowing your child to participate in this study. Your signature below indicates that you have read the information provided above and have decided to allow them to participate in the study. If you later decide that you wish to withdraw your permission for your child to participate in the study you may discontinue his or her participation at any time. You will be given a copy of this document.

| Child's Printed Name: |
|---|
| Printed Name of Parent(s) or Legal Guardian: |
| Signature of Parent(s) or Legal Guardian: |
| Date: |
| For Participants unable to read Witness: I have witnessed the accurate reading of the consent form to the potential participants, and the individual has had the opportunity to ask questions. I confirm that the individual has given consent freely. |
| Witness Name: |
| Witness's Signature / Thumb Print: |
| Date: |
| Signature of Principal/Co- Investigator: Date: |
| Signature of the person obtaining consent: Date: |

# **Informed Consent for Pre- Intervention Focus Group Discussion of Teachers**



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of<br>Health's Fogarty International Center<br>(FIC) in collaboration with Dept of<br>Medicine, Aga Khan University,<br>Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan<br>University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 9. Dr. Aysha Almas 10. Dr. Zainab Samad 11. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. PURPOSE OF THIS PROJECT

You have been invited to participate in a focus group discussion as part of the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors

The purpose of the FGD is to explore participants' views regarding the barriers and facilitators associated with implementing the school-based eHealth NCD prevention program in schools. Furthermore, the participants' viewpoints on the content and design of the program will also be explored.

#### 2. PROCEDURES

The group discussion will be conducted at a secure and comfortable space within the school premises, such as a school library or study room with 6 to 8 other teachers. This discussion will be guided by your experiences, perceptions, and suggestions. A team of two members will conduct this discussion, one will moderate the session, and

the other will record the responses, both in writing and by audio recorder. The group discussion will take about 45 minutes

#### 3. POSSIBLE RISKS OR DISCOMFORT

We do not anticipate any risk or discomfort to you. However, you may decide not to respond to any probes if you feel they are too personal or if talking about them makes you uncomfortable.

#### 4. POSSIBLE BENEFITS

Your active participation in the group discussions will enable us to gain insights into your perspectives on the challenges and facilitators involved in implementing the School-based eHealth NCD prevention program in Pakistani schools. Additionally, these discussions will help us design and develop culturally tailored content for the video sessions and features of the eHealth application.

#### 5. FINANCIAL CONSIDERATIONS

You will be provided meal and travel allowance (if applicable) to participate in the FGD.

#### 6. CONFIDENTIALITY

All information that you provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your personal details. However, any information obtained as a result of your participation in the project may be inspected by the sponsor or by AKU ERC members.

#### 7. TERMINATION OF PROJECT

You are free to choose whether to participate in this project. There will be no penalty or loss of benefits to which you are otherwise entitled if you choose not to participate.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### **AUTHORIZATION**

I have read and understood this consent form, and I volunteer to participate in group-discussion as part of School-based eHealth NCD Prevention Program. I understand that I will receive a copy of this form. I voluntarily choose to participate, but I understand that my consent does not take away any legal rights in the case of negligence or other legal faults of anyone who is involved in this project.

| Name of participant (Printed or Typed): Date: |
|---------------------------------------------------|
| Signature/Thumb Impression of participant : Date: |
| Name of witness (Printed or Typed):<br>Date: |
| Signature/Thumb Impression of the witness: Date: |
| Signature of Principal/Co- Investigator:<br>Date: |
| Signature of the person obtaining consent: Date: |

## **Key Informant Interview**

# **Informed Consent for Pre- Intervention Key Informant Interview - Administrators**



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of<br>Health's Fogarty International Center<br>(FIC) in collaboration with Dept of<br>Medicine, Aga Khan University,<br>Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan<br>University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 12. Dr. Aysha Almas 13. Dr. Zainab Samad 14. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. PURPOSE OF THIS PROJECT

You are being asked to participate in an interview as part of the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors.

The purpose of the KII is to explore participant's views regarding the barriers and facilitators associated with implementing the school-based eHealth NCD prevention program in schools. Furthermore, the participant's viewpoints on the content and design of the program will also be explored.

#### 2. PROCEDURES

The interview will take place at a suitable place within the educational institute facility or the Department of Education, based on your comfort and preference. The prime importance will be given to the place where the participant is comfortable and his/her privacy is ensured.

An interviewer will have a conversation with you regarding your views Another person will be recording your responses, both in writing and by audio recorder. The interview will take about 30 minutes.

#### 3. POSSIBLE RISKS OR DISCOMFORT

We do not anticipate any risk or discomfort to you. However, you may decide not to respond to any question if you feel they are too personal or if talking about them makes you uncomfortable.

#### 4. POSSIBLE BENEFITS

Your active participation in the interview will enable us to gain insights into your perspectives on the challenges and facilitators involved in implementing the Schoolbased eHealth NCD prevention program in Pakistani schools. Additionally, the interview will help us design and develop culturally tailored content for the video sessions and features of the eHealth application.

#### 5. FINANCIAL CONSIDERATIONS

You will be provided meal and travel allowance (if applicable) to participate in the interview

#### 6. CONFIDENTIALITY

All information that you provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your personal details. However, any information obtained as a result of your participation in the project may be inspected by the sponsor or by AKU ERC members.

#### 7. TERMINATION OF PROJECT

You are free to choose whether or not to participate in this project. There are no added benefits or loss of any incentive for your participation in this interview.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### **AUTHORIZATION**

I have read and understood this consent form, and I volunteer to give interview as KII in School-based eHealth NCD Prevention Program. I understand that I will receive a copy of this form. I voluntarily choose to participate, but I understand that my consent does not take away any legal rights in the case of negligence or other legal faults of anyone who is involved in this project.

| Name of participant (Printed or Typed): Date: |
|---------------------------------------------------|
| Signature/Thumb Impression of participant : Date: |
| Name of witness (Printed or Typed):<br>Date: |
| Signature/Thumb Impression of the witness: Date: |
| Signature of Principal/Co- Investigator:<br>Date: |
| Signature of the person obtaining consent: Date: |

## Informed Consent for Pre-Intervention Key Informant Interview – Parent or Guardian



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of<br>Health's Fogarty International Center<br>(FIC) in collaboration with Dept of<br>Medicine, Aga Khan University,<br>Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan<br>University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 15. Dr. Aysha Almas 16. Dr. Zainab Samad 17. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. PURPOSE OF THIS PROJECT

You are being asked to participate in an interview as part of the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors.

The purpose of the KII is to explore participant's views regarding the barriers and facilitators associated with implementing the school-based eHealth NCD prevention program in schools. Furthermore, the participant's viewpoints on the content and design of the program will also be explored.

#### 2. PROCEDURES

The interview will be conducted at a place that is convenient and comfortable for you, whether it is within the educational institute facility, your home, or your office. The prime importance will be given to the place where the participant is comfortable and his/her privacy is ensured.

An interviewer will have a conversation with you regarding your views Another person will be recording your responses, both in writing and by audio recorder. The interview will take about 30 minutes.

#### 3. POSSIBLE RISKS OR DISCOMFORT

We do not anticipate any risk or discomfort to you. However, you may decide not to respond to any question if you feel they are too personal or if talking about them makes you uncomfortable.

#### 4. POSSIBLE BENEFITS

Your active participation in the interview will enable us to gain insights into your perspectives on the challenges and facilitators involved in implementing the School-based eHealth NCD prevention program in Pakistani schools. Additionally, the interview will help us design and develop culturally tailored content for the video sessions and features of the eHealth application.

#### 5. FINANCIAL CONSIDERATIONS

You will be provided meal and travel allowance (if applicable) to participate in the interview.

#### 6. CONFIDENTIALITY

All information that you provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your personal details. However, any information obtained as a result of your participation in the project may be inspected by the sponsor or by AKU ERC members.

#### 7. TERMINATION OF PROJECT

You are free to choose whether or not to participate in this project. There are no added benefits or loss of any incentive for your participation in this interview.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### **AUTHORIZATION**

I have read and understood this consent form, and I volunteer to give interview as KII in School-based eHealth NCD Prevention Program. I understand that I will receive a copy of this form. I voluntarily choose to participate, but I understand that my consent does not take away any legal rights in the case of negligence or other legal faults of anyone who is involved in this project.

| Name of participant (Printed or Typed):<br>Date: |
|---------------------------------------------------|
| Signature/Thumb Impression of participant : Date: |
| Name of witness (Printed or Typed):<br>Date: |
| Signature/Thumb Impression of the witness: Date: |
| Signature of Principal/Co- Investigator:<br>Date: |
| Signature of the person obtaining consent: Date: |

## Intervention

# Assent Form for Students for interventional study (School based eHealth NCD Prevention Program)



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of Health's Fogarty International Centre (FIC) in collaboration with Dept of Medicine, Aga Khan University, Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 18. Dr. Aysha Almas 19. Dr. Zainab Samad 20. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. PURPOSE OF THIS PROJECT

You have been invited to participate in the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors. Based on your eligibility, we invite you to take part in the eHealth education intervention. As part of this study, your school will be randomly assigned to either the intervention or control group. The intervention group will receive health education sessions delivered through multimedia resources in your classrooms, while the control group will follow the standard curriculum. For intervention group, A trained facilitator will guide the sessions, utilizing health education videos during the intervention group sessions. The intervention will last for 2 months, with three sessions per month, each lasting 30 to 40 minutes.

#### 2. PROCEDURES

- If you agree to participate, you will be randomly assigned to either the intervention or control group.
- If you are in intervention group, you will be involved in health education sessions facilitated through a digital application, accessible through internet browsers, including within the school campus if needed. The sessions will include the presentation of health education videos utilizing multimedia. Each session will include 25 to 30 students, and trained facilitators will guide discussions during the sessions.
- If you are in the control group, you will continue with the standard curriculum during the same period.

#### 3. POSSIBLE RISKS OR DISCOMFORT

Your participation in this study or intervention no direct risks or discomforts for you. However, whenever you feel like not participating in the study or intervention you can request for a pause or termination of the study.

#### 4. POSSIBLE BENEFITS

Participating in the eHealth education intervention may help you become more aware of how to prevent non-communicable diseases (NCDs). Furthermore, your participation in this project will assist us in understanding the importance of providing health education on NCDs prevention specifically for Pakistani adolescents. The proposed work has the potential to contribute to the development of effective and culturally appropriate eHealth interventions. It may also contribute to a better understanding of implementation challenges and facilitators in this context. The research outcomes may help shape future strategies for adolescent health, aiming to reduce the burden of NCDs among adolescents and promote healthier lifestyles.

#### 5. FINANCIAL CONSIDERATIONS

You will not be provided any financial incentive to take part in the project.

#### 6. CONFIDENTIALITY

Your responses will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your personal details. However, any information obtained as a result of your participation in the project may be inspected by the sponsor or by AKU ERC members.

#### 7. TERMINATION OF PROJECT

You are free to choose whether to participate in this project. There are no added benefit or loss of any incentive with regard to your participation in the project. You will be provided with any significant new findings developed during this study that may relate to or influence your willingness to continue participation. Please inform the facilitator if you wish to terminate your participation in the project.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### **AUTHORIZATION**

I have read and understood this consent form, and I volunteer to participate in this project. I understand that I will receive a copy of this form. I voluntarily choose to participate, but I understand that my consent does not take away any legal rights in the case of negligence or other legal faults of anyone who is involved in this project.

Name of participant (Printed or Typed):

Date:

Signature / Thumb Impression of participant:

Date:

Signature of Principal/Co- Investigator:

Date:

Signature of the person obtaining consent:

Date:

## Consent Form from Parents for their child participation in interventional study (School based eHealth NCD Prevention Program)



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of Health's Fogarty International Center (FIC) in collaboration with Dept of Medicine, Aga Khan University, Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 21. Dr. Aysha Almas 22. Dr. Zainab Samad 23. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. Introduction

The purpose of this form is to provide you (as the parent of a prospective research study participant) information that may affect your decision as to whether or not to let your child participate in this research study. The person performing the research will describe the study to you and answer all your questions. Read the information below and ask any questions you might have before deciding whether or not to give your permission for your child to take part. If you decide to let your child participate in this study, this form will be used to record your permission.

#### 2. PURPOSE OF THIS PROJECT

If you agree, your child will be asked to participate in the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors.

Based on your child's eligibility, we invite your child to take part in the eHealth education intervention. As part of this study, your child's school will be randomly assigned to either the intervention or control group. The intervention group will receive

health education sessions delivered through multimedia resources in your classrooms, while the control group will follow the standard curriculum. For intervention group, A trained facilitator will guide the sessions, utilizing health education videos during the intervention group sessions. The intervention will last for 2 months, with three sessions per month, each lasting 30 to 40 minutes.

#### 3. PROCEDURES

- If you agree to participate, your child will be randomly assigned to either the intervention or control group.
- If your child is in intervention group, your child will be involved in health education sessions facilitated through a digital application, accessible through internet browsers, including within the school campus if needed. The sessions will include the presentation of health education videos utilizing multimedia. Each session will include 25 to 30 students, and trained facilitators will guide discussions during the sessions.
- If you child is in the control group, your child will continue with the standard curriculum during the same period.

#### 4. POSSIBLE RISKS OR DISCOMFORT

Your child participation in receiving eHealth education intervention poses no direct risks or discomforts for her/him. However, whenever your child feel like not participating in the session, your child can request for a pause or termination of session.

#### 5. POSSIBLE BENEFITS

Your child's active participation in the eHealth education intervention may help your child become more aware of how to prevent non-communicable diseases (NCDs). Furthermore, your child participation in this project will assist us in understanding the importance of providing health education on NCDs prevention specifically for Pakistani adolescents. The proposed work has the potential to contribute to the development of effective and culturally appropriate eHealth interventions. It may also contribute to a better understanding of implementation challenges and facilitators in this context. The research outcomes may help shape future strategies for adolescent health, aiming to reduce the burden of NCDs among adolescents and promote healthier lifestyles.

#### 6. FINANCIAL CONSIDERATIONS

Neither you nor your child will receive any type of payment participating in this study.

#### 7. CONFIDENTIALITY

Your child's privacy and the confidentiality of his/her data will be protected by keeping all information that your child provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your child's personal details. Your child's research records will not be released without your consent unless required by law or a court order. If it becomes necessary for the Ethics Review Committee to review the study records, information that can be linked to your child will be protected to the extent permitted by law. The data resulting from your child's participation may be made available to other researchers in the future for research purposes without identification. In these cases, the data will contain no identifying information that could associate it with your child, or with your child's participation in any study.

#### 8. TERMINATION OF PROJECT

Your child's participation in this study is voluntary. Your child may decline to participate or to withdraw from participation at any time. Withdrawal or refusing to participate will not affect their treatment/procedure or relationship with Aga Khan University in anyway. You can agree to allow your child to be in the study now and change your mind later without any penalty.

In addition to your permission, your child must agree to participate in the study. If your child does not want to participate they will not be included in the study and there will be no penalty. If your child initially agrees to be in the study s/he can change their mind later without any penalty.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### **AUTHORIZATION**

You are making a decision about allowing your child to participate in this study. Your signature below indicates that you have read the information provided above and have decided to allow them to participate in the study. If you later decide that you wish to withdraw your permission for your child to participate in the study you may discontinue his or her participation at any time. You will be given a copy of this document.

| Child's Printed Name: |
|---|
| Printed Name of Parent(s) or Legal Guardian: |
| Signature of Parent(s) or Legal Guardian: |
| Date: |
| For Participants unable to read Witness: I have witnessed the accurate reading of the consent form to the potential participants, and the individual has had the opportunity to ask questions. I confirm that the individual has given consent freely. |
| Witness Name: |
| Witness's Signature / Thumb Print: |
| Date: |
| Signature of Principal/Co- Investigator: Date: |
| Signature of the person obtaining consent: Date: |

## **Post Intervention**

# **Assent Form for Post-Intervention Focus Group Discussion of Students**



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness in<br>Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of Health's Fogarty International Center (FIC) in collaboration with Dept of Medicine, Aga Khan University, Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 24. Dr. Aysha Almas 25. Dr. Zainab Samad 26. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. PURPOSE OF THIS PROJECT

You have been invited to participate in a focus group discussion as part of the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors.

The purpose of the FGD is to explore the perceptions of participants regarding the usefulness, acceptability, and task technology fitness of a school-based eHealth NCD prevention program in improving the knowledge, attitudes, and practices of adolescents.

#### 2. PROCEDURES

The group discussion will be conducted at a secure and comfortable space within the school premises, such as a school library or study room with 6 to 8 other students. This discussion will be guided by your experiences, perceptions, and suggestions. A team of two members will conduct this discussion, one will moderate the session, and the other will record the responses, both in writing and by audio recorder. The group discussion will take about 45 minutes

#### 3. POSSIBLE RISKS OR DISCOMFORT

We do not anticipate any risk or discomfort to you. However, you may decide not to respond to any probes if you feel they are too personal or if talking about them makes you uncomfortable.

#### 4. POSSIBLE BENEFITS

By actively participating in the group discussions, you will provide valuable insights on the school-based eHealth NCD prevention program's usefulness, acceptability, and task technology fitness. Your input will play a crucial role in shaping future eHealth interventions and refining the eHealth app's interface and content.

Your contribution will help us better understand how effective and user-friendly the program was in increasing NCDs prevention awareness among adolescents. Additionally, your input will assist us in identifying ways to further improve the program's effectiveness and user-friendliness

#### 5. FINANCIAL CONSIDERATIONS

You will be provided meal & travel allowance (if applicable) to participate in the FGD.

#### 6. CONFIDENTIALITY

All information that you provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your personal details. However, any information obtained as a result of your participation in the project may be inspected by the sponsor or by AKU ERC members.

#### 7. TERMINATION OF PROJECT

You are free to choose whether to participate in this project. There will be no penalty or loss of benefits to which you are otherwise entitled, if you choose not to participate.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### **AUTHORIZATION**

I have read and understood this form, and I volunteer to participate in group-discussion as part of School-based eHealth NCD Prevention Program. I understand that I will receive a copy of this form. I voluntarily choose to participate, but I understand that my consent does not take away any legal rights in the case of negligence or other legal faults of anyone who is involved in this project.

| Name of participant (Printed or Typed):<br>Date: |
|---------------------------------------------------|
| Signature/Thumb Impression of participant : Date: |
| Name of witness (Printed or Typed):<br>Date: |
| Signature/Thumb Impression of the witness: |

| Signature of Principal/Co- Investigator: Date: |
|-------------------------------------------------|
| Signature of the person obtaining consent Date: |

## Consent Form for Post-Intervention Focus Group Discussion of Students



| Project Information | |
|---|---|
| Project Title: School-based eHealth NCD<br>Prevention Program to Improve Awareness<br>in Adolescents from Urban Pakistan | Project ID: |
| ERC Ref No: | Sponsor: National Institutes of Health's Fogarty International Center (FIC) in collaboration with Dept of Medicine, Aga Khan University, Karachi, Pakistan |
| Principal Investigator: Dr. Tazeen Saeed Ali | Organization: The Aga Khan<br>University |
| Location: Karachi | Phone: +92 21 3493 0051 Ext. 5400 |
| Other Investigators: 27. Dr. Aysha Almas 28. Dr. Zainab Samad 29. Muhammad Shahid Khan | Organization:<br>The Aga Khan University |
| Location: Karachi, Pakistan | Phone: +92 21 3414 6880 |

#### 1. Introduction

The purpose of this form is to provide you (as the parent of a prospective research study participant) information that may affect your decision as to whether or not to let your child participate in this research study. The person performing the research will describe the study to you and answer all your questions. Read the information below and ask any questions you might have before deciding whether or not to give your permission for your child to take part. If you decide to let your child participate in this study, this form will be used to record your permission.

#### 2. PURPOSE OF THIS PROJECT

If you agree, your child will be asked to participate in a focus group discussion as part of the School-based eHealth NCD Prevention Program, which aims to enhance the knowledge, attitude, and practices of adolescents regarding NCD prevention, specifically in terms of diet, physical activity, and other related factors.

The purpose of the FGD is to explore the perceptions of participants regarding the usefulness, acceptability, and task technology fitness of a school-based eHealth NCD

prevention program in improving the knowledge, attitudes, and practices of adolescents.

#### 3. PROCEDURES

The group discussion will be conducted at a secure and comfortable space within the school premises, such as a school library or study room with 6 to 8 other students. This discussion will be guided by your child's experiences, perceptions, and suggestions. A team of two members will conduct this discussion, one will moderate the session, and the other will record the responses, both in writing and by audio recorder. The group discussion will take about 45 minutes.

#### POSSIBLE RISKS OR DISCOMFORT

We do not anticipate any risk or discomfort to the participant. However, your child may decide not to respond to any probes if s/he feel they are too personal or if talking about them makes him/her uncomfortable.

#### 4. POSSIBLE BENEFITS

Your child's active participation in the group discussions will enable us to gain insights on the on the school-based eHealth NCD prevention program's usefulness, acceptability, and task technology fitness. Your child input will play a crucial role in shaping future eHealth interventions and refining the eHealth app's interface and content.

Your child contribution will help us better understand how effective and user-friendly the program was in increasing NCDs prevention awareness among adolescents. Additionally, your child input will assist us in identifying ways to further improve the program's effectiveness and user-friendliness.

#### 5. FINANCIAL CONSIDERATIONS

Your child will be provided meal and travel allowance (if applicable) to participate in the FGD.

#### 6. CONFIDENTIALITY

Your child's privacy and the confidentiality of his/her data will be protected by keeping all information that your child provide will be kept confidential. The analysis will be done at a group level. Only the primary research team will be aware of your child's personal details. Your child's research records will not be released without your consent unless required by law or a court order. If it becomes necessary for the Ethics Review Committee to review the study records, information that can be linked to your child will be protected to the extent permitted by law. The data resulting from your child's participation may be made available to other researchers in the future for research purposes without identification. In these cases, the data will contain no identifying information that could associate it with your child, or with your child's participation in any study.

#### 7. TERMINATION OF PROJECT

Your child's participation in this study is voluntary. Your child may decline to participate or to withdraw from participation at any time. Withdrawal or refusing to participate will not affect their treatment/procedure or relationship with Aga Khan University in anyway. You can agree to allow your child to be in the study now and

change your mind later without any penalty. In addition to your permission, your child must agree to participate in the study. If your child does not want to participate they will not be included in the study and there will be no penalty. If your child initially agrees to be in the study s/he can change their mind later without any penalty.

#### 8. AVAILABLE SOURCES OF INFORMATION

Any further questions you have about this project will be answered by the

Investigator: Dr. Tazeen Saeed Ali

Phone Number: +92 21 3493 0051 Ext. 5400

#### 9. AUTHORIZATION

You are making a decision about allowing your child to participate in this study. Your signature below indicates that you have read the information provided above and have decided to allow them to participate in the study. If you later decide that you wish to withdraw your permission for your child to participate in the study, you may discontinue his or her participation at any time. You will be given a copy of this document.

| document. |
|---|
| Child's Printed Name: |
| Printed Name of Parent(s) or Legal Guardian: |
| Signature of Parent(s) or Legal Guardian: |
| Date: |
| For Participants unable to read Witness: I have witnessed the accurate reading of the consent form to the potential participants, and the individual has had the opportunity to ask questions. I confirm that the individual has given consent freely. |
| Witness Name: |
| Witness's Signature / Thumb Print: |
| Date: |
| Signature of Principal/Co- Investigator: |
| Date: |
| Signature of the person obtaining consent: |
| Date: |